CLINICAL TRIAL: NCT02174900
Title: Evaluation of the Safety of Primaquine in Combination With Artemether-lumefantrine in Glucose-6-phosphate Dehydrogynase Deficient Males With an Asymptomatic Malaria Infection in Burkina Faso (SAFEPRIM)
Brief Title: Safety of Primaquine + Artemether-lumefantrine in G6PD Deficient Males With an Asymptomatic Malaria Infection (SAFEPRIM)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Centre national de recherche et de formation sur le paludisme (Other Government); University Medical Center Nijmegen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFEPRIM
Record Dates: First submitted 2014-06-11; First posted 2014-06-26 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Malaria
Keywords: G6PD deficiency; safety; transmission
MeSH Terms: conditions — Malaria; Glucosephosphate Dehydrogenase Deficiency | interventions — Artemether, Lumefantrine Drug Combination; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- G6PD deficient 0.25 mg/kg PQ + AL (Experimental): G6PD deficient males receiving Artemether-Lumefantrine (AL) + 0.25 mg/kg primaquine
  Interventions: Drug: Artemether-Lumefantrine (AL) + 0.25 mg/kg primaquine
- G6PD deficient receiving AL only (Active Comparator): G6PD deficient males receiving Artemether-Lumefantrine (AL) combination
  Interventions: Drug: Artemether-Lumefantrine (AL) combination
- G6PD normal 0.25 mg/kg PQ + AL (Active Comparator): G6PD normal males receiving Artemether-Lumefantrine (AL) + 0.25 mg/kg primaquine
  Interventions: Drug: Artemether-Lumefantrine (AL) + 0.25 mg/kg primaquine
- G6PD normal 0.4 mg/kg PQ + AL (Active Comparator): G6PD normal males receiving Artemether-Lumefantrine (AL) + 0.4 mg/kg primaquine
  Interventions: Drug: Artemether-Lumefantrine (AL) + 0.4 mg/kg primaquine
- G6PD-deficient 0.4 mg/kg PQ + AL (Experimental): G6PD deficient males receiving Artemether-Lumefantrine (AL) + 0.4 mg/kg primaquine
  Interventions: Drug: Artemether-Lumefantrine (AL) + 0.4 mg/kg primaquine

INTERVENTIONS:
Drug: Artemether-Lumefantrine (AL) + 0.25 mg/kg primaquine
  Arms: G6PD deficient 0.25 mg/kg PQ + AL; G6PD normal 0.25 mg/kg PQ + AL
Drug: Artemether-Lumefantrine (AL) combination
  Arms: G6PD deficient receiving AL only
Drug: Artemether-Lumefantrine (AL) + 0.4 mg/kg primaquine
  Arms: G6PD normal 0.4 mg/kg PQ + AL; G6PD-deficient 0.4 mg/kg PQ + AL

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of increasing doses of primaquine in combination with artemether-lumefantrine in G6PD deficient males with an asymptomatic P. falciparum malaria infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male gender
2. Age ≥18 years and ≤45 years
3. BMI ≥16
4. P. falciparum parasitaemia at any density
5. G6PD deficiency by Beutler Fluorescent Spot test for intervention groups and control group receiving AL only (N=50)
6. G6PD normal activity by Beutler Fluorescent Spot test for control groups (N=20)
7. Informed consent by participant

Exclusion Criteria:

1. Enrolled in another clinical trial
2. Fever >37.5°C (tympanic) or history of fever in the last 24 hours
3. Evidence of severe illness / danger signs or active infection other than malaria
4. Known allergy to study medications
5. Hb <11 g/dL
6. Antimalarials taken within the last 2 weeks
7. PQ taken within the last 4 weeks and blood transfusion within the last 90 days
8. Non-falciparum malaria co-infection
9. Current use of tuberculosis or anti-retroviral medication, sulphonamides, dapsone, nitrofurantoin, , nalidixic acid, ciprofloxacin, , methylene blue, toluidine blue phenazopyridine and co-trimoxazole.
10. History of severe chronic illness

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Haemoglobin concentration relative to baseline value | 28 days
  Haemoglobin concentration relative to baseline value

SECONDARY OUTCOMES:
Gametocyte clearance time | 14 days
  Gametocyte clearance time

CONTACTS AND LOCATIONS:
Overall Officials: Teun Bousema, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Burkina Faso

REFERENCES:
- [Derived] Bastiaens GJH, Tiono AB, Okebe J, Pett HE, Coulibaly SA, Goncalves BP, Affara M, Ouedraogo A, Bougouma EC, Sanou GS, Nebie I, Bradley J, Lanke KHW, Niemi M, Sirima SB, d'Alessandro U, Bousema T, Drakeley C. Safety of single low-dose primaquine in glucose-6-phosphate dehydrogenase deficient falciparum-infected African males: Two open-label, randomized, safety trials. PLoS One. 2018 Jan 11;13(1):e0190272. doi: 10.1371/journal.pone.0190272. eCollection 2018. PMID 29324864